CLINICAL TRIAL: NCT06077149
Title: A Comparison of Immunogenicity of Licensed RSV Vaccines in Residents of Long-Term Care Facilities (LTCF) to Community-dwelling Older Adults
Brief Title: Immunogenicity of RSV Vaccines in Residents of Long-Term Care Facilities (LTCF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ann Falsey, Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00008699
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Laboratory testing will be blinded to vaccine and study cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long-term care facility residents (Experimental): Licensed RSV vaccine IM x 1. Specific product to be determined availability at the facility as SOC
  Interventions: Biological: RSV vaccine
- community dwelling adults (Active Comparator): Licensed RSV vaccine IM x1. The proportion of specific products will be matched to the LTCF cohort
  Interventions: Biological: RSV vaccine

INTERVENTIONS:
Biological: RSV vaccine — All participants will get either the Pfizer RSV vaccine (RSVpreF (ABRYSVO)) or the GSK RSV vaccine (RSVpreF (AREXVY)) at 120 ug of the RSV prefusion F antigen intramuscularly in the the non-dominant deltoid muscle.
  Long-term care facility residents will get whichever vaccine is available at the facility as part of standard of care. Community cohort will be matched proportionally

SUMMARY:
This clinical trial is studying the newly licensed RSV vaccines in adults over age 60 years living in long-term care facilities (nursing homes) by comparing the immune response to their vaccine to adults over age 60 years living in the community.

DETAILED DESCRIPTION:
This was an open label non-inferiority study to evaluate immunogenicity where all participants received either the Pfizer RSV Vaccine (ABRYSVO) or GSK RSV Vaccine (AREXVY) as part of Standard of Care (SOC). Hereafter, vaccines will be referred to as Pfizer and GSK.

The study was conducted at the University of Rochester Medical Center (URMC) Infectious Disease Research Clinic (IDRC) and 2 local LTCFs. Vaccinations were carried out between November and December 2023. LTCF A provided GSK vaccine and LTCF B provided Pfizer vaccine to their residents as part of SOC. The community cohort was divided equally to receive Pfizer and GSK to mirror the Pfizer and GSK vaccinations in LTCF. The study was reviewed and approved by the University of Rochester Institutional Review Board and leadership at the local LTCFs. Participants or their legally authorized representative (LAR) signed written informed consent. Verbal consent by LAR was also accepted given the minimal risk nature of the study.

Participants:

Inclusion criteria were intended to be broad with relatively few exclusions to reflect a real-life population in LTCF and the older adults in the community. Inclusion criteria included: ≥60 years of age living LTCF or residing independently in the community, planning to receive a SOC RSV vaccine, life expectancy of >6 months, able to sign informed consent or to provide consent via a LAR. Exclusions included: history of a current immunosuppressive condition or medications, history of hypersensitivity or reaction to any vaccine component, any routine vaccination within a 14-day window before or planned after RSV vaccination, previous receipt or intended receipt of an RSV vaccine outside the study, receipt of blood/plasma products or immunoglobulin within 60 days before RSV vaccination, and documented RSV infection within 2 months prior to enrollment.

Study Procedures:

Prior to any study procedures informed consent was obtained from the participant or LAR. At enrollment demographic and medical history data were collected. A clinical assessment including vital signs and a symptom directed targeted physical exam was performed. Ten 10cc of blood was collected. Vaccination in LTCF were performed by the staff at each facility per SOC and the vaccine product and date of vaccination recorded. Vaccination of the community cohort was performed in the IDRC at enrollment visit. Visit two was scheduled 28 to 42 days following vaccination at which time a second 10cc blood sample was collected and participants were queried about any intercurrent illnesses. Results of any viral testing performed as part of standard of care were recorded. If a participant had an intercurrent RSV infection prior to RSV vaccination and vaccination was deferred, visit 2 was scheduled 28 -42 days after infection was documented.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age who live in skilled nursing facilities or reside independently in the community
* Life expectancy of >6 months, as assessed by the investigator
* Able to sign informed consent or to provide consent via a legally authorized representative (LAR)

Exclusion Criteria:

* History of a current immunosuppressive condition or receipt of chemotherapy or other immunosuppressive or cytotoxic therapy, including chronic prednisone use of ≥ 20 mg/day for more than 14 days within 3 months of study vaccination
* History of hypersensitivity or reaction to any vaccine component
* Simultaneous administration of another vaccine (influenza, SARS-CoV-2) or within a 14-day window before or after intervention
* Previous receipt or intended receipt of an RSV vaccine outside the study
* Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration.
* Documented RSV infection within 2 months prior to study intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Falsey, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Long-term care facility residents: Licensed RSV vaccine IM x 1. Specific product to be determined availability at the facility as SOC
  RSV vaccine: All participants will get either the Pfizer RSV vaccine (RSVpreF (ABRYSVO)) or the GSK RSV vaccine (RSVpreF (AREXVY)) at 120 ug of the RSV prefusion F antigen intramuscularly in the the non-dominant deltoid muscle.
  Long-term care facility residents will get whichever vaccine is available at the facility as part of standard of care. Community cohort will be matched proportionally
- community dwelling adults: Licensed RSV vaccine IM x1. The proportion of specific products will be matched to the LTCF cohort
  RSV vaccine: All participants will get either the Pfizer RSV vaccine (RSVpreF (ABRYSVO)) or the GSK RSV vaccine (RSVpreF (AREXVY)) at 120 ug of the RSV prefusion F antigen intramuscularly in the the non-dominant deltoid muscle.
  Long-term care facility residents will get whichever vaccine is available at the facility as part of standard of care. Community cohort will be matched proportionally
Period: Overall Study
Arm/Group | Long-term care facility residents | community dwelling adults
Started | 76 | 76
Completed | 70 | 76
Not Completed | 6 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — RSV infection before vaccination | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long-term care facility residents | community dwelling adults | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (9.6) | 72.6 (6.3) | 75.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 72 | 75 | 147
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 69 | 72 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 152
Number of participants with diabetes mellitus [Count of Participants; unit: Participants] | 25 | 16 | 41
Number of participants with coronary artery disease [Count of Participants; unit: Participants] | 28 | 6 | 34
Number of participants with congestive heart failure [Count of Participants; unit: Participants] | 20 | 2 | 22
Number of participants with obstructive pulmonary disease [Count of Participants; unit: Participants] | 5 | 14 | 19
Number of participants with Asthma [Count of Participants; unit: Participants] | 5 | 5 | 10
Number of participants with hypertension [Count of Participants; unit: Participants] | 61 | 27 | 88
Number of participants with chronic kidney disease [Count of Participants; unit: Participants] | 24 | 2 | 26
Number of participants with cerebrovascular accident [Count of Participants; unit: Participants] | 24 | 0 | 24
Number of participants with dementia [Count of Participants; unit: Participants] | 33 | 0 | 33
Number of participants with cancer [Count of Participants; unit: Participants] | 15 | 4 | 19
Mean number of medical conditions [Mean (Standard Deviation); unit: number of medical conditions] | 5.6 (1.8) | 2.2 (1.8) | 3.9 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise Against RSV Fa Protein
Description: Microneutralization Assay (MNA): Serum neutralizing titers will be performed using an established microneutralization method for RSV A and B strains. Briefly, 2-fold serum dilutions are incubated with 75 plaque forming units of RSV for 30 min at room temperature followed by the addition of 104HEp-2cells in 96-well culture plates. After 3 days, the quantity of RSV antigen is determined by enzyme immunoassay using a monoclonal antibody to the RSV Fa protein. The geometric mean fold rise is the neutralizing antibody titer at day 30 divided by the neutralizing antibody titer at day 0. Calculated as the geometric mean of the fold rise (post-vaccination titer divided by baseline titer) across participants.
Time Frame: 30 days
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Long-term care facility residents | community dwelling adults
Number analyzed (Participants) | 70 | 76
fold change | 12.5 [12.0 to 12.9] | 9.9 [9.8 to 9.9]
Statistical Analysis 1: Comparison: Long-term care facility residents vs community dwelling adults; Test type: Non-Inferiority — The primary outcome of the study was to demonstrate the noninferiority in antibody response at 30 days for any RSV vaccine between the LTCF group and the community group. A sample size of 152 participants (76 per group) was expected to provide 80% power to demonstrate noninferiority of 1 month GMT to within a relative noninferiority margin of 1.5-fold using a 1-sided 0.05-level linear model-based t test comparing log (1-month titer) by population, adjusted for vaccine and log (baseline titer); p = 0.14, t-test, 2 sided

2. Primary Outcome: Geometric Mean Fold Rise Against RSV Fb Protein
Description: Microneutralization Assay (MNA): Serum neutralizing titers will be performed using an established microneutralization method for RSV A and B strains. Briefly, 2-fold serum dilutions are incubated with 75 plaque forming units of RSV for 30 min at room temperature followed by the addition of 104HEp-2cells in 96-well culture plates. After 3 days, the quantity of RSV antigen is determined by enzyme immunoassay using a monoclonal antibody to the RSV Fb protein. The geometric mean fold rise is the neutralizing antibody titer at day 30 divided by the neutralizing antibody titer at day 0. Calculated as the geometric mean of the fold rise (post-vaccination titer divided by baseline titer) across participants.
Time Frame: 30 days
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Long-term care facility residents | community dwelling adults
Number analyzed (Participants) | 70 | 76
fold change | 11.0 [10.5 to 11.6] | 8.7 [8.6 to 8.8]
Statistical Analysis 1: Comparison: Long-term care facility residents vs community dwelling adults; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.17, t-test, 2 sided

3. Primary Outcome: Geometric Mean Fold Rise Against RSV A2 Protein
Description: Microneutralization Assay (MNA): Serum neutralizing titers will be performed using an established microneutralization method for RSV A and B strains. Briefly, 2-fold serum dilutions are incubated with 75 plaque forming units of RSV for 30 min at room temperature followed by the addition of 104HEp-2cells in 96-well culture plates. After 3 days, the quantity of RSV antigen is determined by enzyme immunoassay using a monoclonal antibody to the RSV A2 protein. The geometric mean fold rise is the neutralizing antibody titer at day 30 divided by the neutralizing antibody titer at day 0. Calculated as the geometric mean of the fold rise (post-vaccination titer divided by baseline titer) across participants.
Time Frame: 30 days
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Long-term care facility residents | community dwelling adults
Number analyzed (Participants) | 70 | 76
fold change | 15.5 [15.2 to 16.0] | 12.8 [12.6 to 12.9]
Statistical Analysis 1: Comparison: Long-term care facility residents vs community dwelling adults; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.32, t-test, 2 sided

4. Secondary Outcome: Ratio of Fold Response of RSV A2 Titer to Fa Titer
Description: the ratio of fold response of RSV A2 neutralizing titer to Fa IgG binding titers was calculated as a measure of the relative proportion of functional F antibody produced
Time Frame: 30 days
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of A2 to Fa
Arm/Group | Long-term care facility residents | community dwelling adults
Number analyzed (Participants) | 70 | 76
proportion of A2 to Fa | 1.15 [1.00 to 1.32] | 1.18 [1.07 to 1.29]
Statistical Analysis 1: Comparison: Long-term care facility residents vs community dwelling adults; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.82, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Long-term care facility residents | community dwelling adults
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT06077149/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT06077149/ICF_001.pdf